CLINICAL TRIAL: NCT03015636
Title: Better Sleep in Psychiatric Care - ADHD. A Randomized Naturalistic Study of a Psychological Group Treatment for Sleep Problems in Psychiatric Patients With Attention Deficit Hyperactivity Disorder.
Brief Title: Better Sleep in Psychiatric Care - ADHD.
Acronym: BSIP-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Department of ADHD, Northern Stockholm Psychiatry (Unknown)
Responsible Party: Principal Investigator, Susanna Jernelöv, PhD, LP, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1988-31
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Sleep Problem; ADHD
Keywords: Cognitive Behaviour Therapy; Psychological Intervention
MeSH Terms: conditions — Parasomnias; Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral: Adjusted CBT-i for ADHD (Experimental): Cognitive Behavioral group intervention for sleep problems in ADHD, based on Cognitive Behavioral Therapy for insomnia and behavioral treatment for Sleep Phase Disorders.
  Interventions: Behavioral: Adjusted CBT-i for ADHD
- Treatment as Usual (Other): Treatment as Usual. (After about ten weeks, participants in this condition are offered the experimental group treatment.)
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Adjusted CBT-i for ADHD — This is a version of CBT for insomnia (CBT-i) developed during the pilot phase of this Project. Traditional CBT-i is adjusted for use in the adult ADHD population. This behavioral intervention adresses not only traditional aspects of insomnia, but also sleep phase problems and other aspects of sleep specifically relevant to the ADHD-population. Treatment is given as 10 weekly group sessions with telephone calls from the therapist between sessions to increase adherence and adress individual patient needs.
  Arms: Behavioral: Adjusted CBT-i for ADHD
Other: Treatment as Usual — Usual care at the ADHD-clinic. This mostly entails managing pharmacological treatment for ADHD, comorbid psychiatric problems and/or sleep problems. The clinic also provides different group treatments, for instance mindfulness groups and groups for developing behavioral strategies for managing ADHD symptoms, and individual therapy.
  Arms: Treatment as Usual

SUMMARY:
Cognitive Behavioral Therapy (CBT) is treatment of choice for insomnia (CBT-i). Many patients in psychiatric care have sleep problems including insomnia, but are rarely given the choice to participate in CBT to improve their sleep. Patients with ADHD is a patient group with high levels of sleep difficulties. Sleep problems in this patient group can be both more general such as insomnia, but can also be related to the ADHD itself and to the use of ADHD medication. In a previous pilot study, the investigators developed a version of CBT-i that would target sleep problems in this population. The basis was CBT-i, but with more emphasis on sleep promoting behaviors specific to ADHD (e.g. appropriate timing of ADHD-medication), techniques that would also alleviate sleep phase problems, (e.g. the systematic use of light and darkness), and techniques to target more general sleep disturbing habits (e.g. not winding down before bed time), that are also common in patients with ADHD. This treatment was well tolerated and gave moderate effects on insomnia severity in the pilot study. In a naturalistic randomized controlled trial, the investigators now evaluate the effects of this psychological treatment on sleep and symptoms of ADHD in patients at the ADHD-clinics, Northern Stockholm Psychiatry, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient at the ADHD-clinics Northern Stockholm Psychiatry
* Experiencing sleep problems (subjective report)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-12; Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Changes from base-line to 10 weeks and 3 months
  7-item, self-rated questionnaire measuring change in insomnia severity.

SECONDARY OUTCOMES:
Actigraphy | Continuously from treatment start (week 1) to the last week of treatment (week 10)
  An actigraph is placed on the participant's arm for one week. It measures participants' activity in the form of movements. It can be used for acquiring data on sleep and daytime activity, including calculated sleep latency, total sleep time, sleep efficiency, wake after sleep onset, variability in sleep timing and daytime activity.
Sleep diary | Changes from base-line to 10 weeks and 3 months
  Daily self-ratings on a number of sleep parameters, resulting in several measures including sleep latency, wake after sleep onset, total sleep time, sleep efficiency, subjective sleep quality and variability in sleep timing

OTHER OUTCOMES:
Brunnsviken brief quality of life scale | Changes from base-line to 10 weeks and 3 months
  12-items self-rating questionnaire measuring quality of life.
Adult ADHD Self-Report Scale | Changes from base-line to 10 weeks and 3 months
  18-items self-report questionnaire measuring ADHD-symptoms.
Dysfunctional Beliefs and Attitudes about Sleep | Changes from base-line to 10 weeks and 3 months
  10-items self-rating questionnaire measuring sleep related cognitions.
Sleep Problems Acceptance Questionnaire | Changes from base-line to 10 weeks and 3 months
  8-items self-rating questionnaire measuring acceptance of sleep problems.
Sleep habits and behaviors | Changes from base-line to 10 weeks and 3 months
  Self-rating questionnaire regarding the use of sleep promoting behaviors. The questionnaire was constructed for the current project and consists of two parts. The first part includes 16 statements such as "Last week I got out of bed within 15 minutes of waking up" to be answered by number of days the last week this was true (i.e. from 0 to 7). The other part is to be answered on a 6-point Likert scale from "Not at all true" to "Entirely true", with 7 statements like "I get out of bed the same time every morning".

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, LP, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of ADHD, Northern Stockholm Psychiatry, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Lindner P, Frykheden O, Forsstrom D, Andersson E, Ljotsson B, Hedman E, Andersson G, Carlbring P. The Brunnsviken Brief Quality of Life Scale (BBQ): Development and Psychometric Evaluation. Cogn Behav Ther. 2016 Apr;45(3):182-95. doi: 10.1080/16506073.2016.1143526. Epub 2016 Feb 17. PMID 26886248
- [Background] Adler LA, Spencer T, Faraone SV, Kessler RC, Howes MJ, Biederman J, Secnik K. Validity of pilot Adult ADHD Self- Report Scale (ASRS) to Rate Adult ADHD symptoms. Ann Clin Psychiatry. 2006 Jul-Sep;18(3):145-8. doi: 10.1080/10401230600801077. PMID 16923651
- [Background] Espie CA, Inglis SJ, Harvey L, Tessier S. Insomniacs' attributions. psychometric properties of the Dysfunctional Beliefs and Attitudes about Sleep Scale and the Sleep Disturbance Questionnaire. J Psychosom Res. 2000 Feb;48(2):141-8. doi: 10.1016/s0022-3999(99)00090-2. PMID 10719130
- [Background] Bothelius K, Jernelov S, Fredrikson M, McCracken LM, Kaldo V. Measuring Acceptance of Sleep Difficulties: The Development of the Sleep Problem Acceptance Questionnaire. Sleep. 2015 Nov 1;38(11):1815-22. doi: 10.5665/sleep.5170. PMID 26085302